CLINICAL TRIAL: NCT04911491
Title: Inspiratory Muscle Strength Training for Lowering Systolic Blood Pressure in Midlife and Older Adults With Chronic Kidney Disease
Brief Title: Inspiratory Muscle Strength Training in Chronic Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-3000; R01DK130255 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-06-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases; Hypertension; Aging; Blood Pressure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IMST (Experimental): This group will perform high-resistance (75% of maximal inspiratory pressure) inspiratory muscle strength training (IMST), 30 inhalations/session, 6 days/week.
  Interventions: Device: IMST
- Control (Sham Comparator): This group will perform low-resistance (15% of maximal inspiratory pressure) inspiratory muscle strength training, 30 inhalations/session, 6 days/week.
  Interventions: Device: Sham Training

INTERVENTIONS:
Device: IMST — Inspiratory muscle strength training (IMST) is a form of physical training that utilizes the diaphragm and accessory respiratory muscles to repeatedly inhale against resistance using a handheld device.
  Arms: IMST
Device: Sham Training — Repeated inhalations against a low resistance will be performed using a handheld device.
  Arms: Control

SUMMARY:
More than 80% of individuals with chronic kidney disease have concomitant hypertension and the majority fail to achieve blood pressure control <130/80 mmHg, leading to high risk of cardiovascular diseases and end-stage kidney disease. A stepwise combination of lifestyle modifications and drug therapy is recommended to lower blood pressure; however, adherence to time-intensive lifestyle interventions such as aerobic exercise in patients with chronic kidney disease is poor. This clinical trial seeks to establish the efficacy of high-resistance inspiratory muscle strength training, a novel time-efficient lifestyle intervention, for lowering systolic blood pressure and improving endothelial function in midlife and older adults with moderate-to-severe chronic kidney disease and inadequately controlled hypertension, and to use innovate translational assessments to understand the mechanisms involved.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major public health concern that has reached epidemic proportions. Hypertension is a leading modifiable risk factor for cardiovascular disease (CVD) and end-stage kidney disease, yet 50-70% of adults with CKD fail to achieve blood pressure (BP) control to <130/80 mmHg. A key process linking high systolic BP (SBP) to CVD is vascular endothelial dysfunction, which is due in part to increased reactive oxygen species and decreased nitric oxide. Nitric oxide is also critical in the regulation of renal blood flow, which is intimately related to blood pressure and vascular function. High-resistance inspiratory muscle strength training (IMST) is a novel lifestyle intervention involving repeated inhalations against a resistive load using a hand-held device. This study will test whether high-resistance IMST (75% of maximal inspiratory pressure [75% PImax]; 30 breaths [5 min]/day, 6 days [30 min]/week) vs. Sham training (15% PImax) reduces resting systolic blood pressure in midlife and older adults (>50 years) with moderate-to-severe CKD and inadequately controlled hypertension. Changes in 24-hr systolic blood pressure and endothelial function (brachial artery flow-mediated dilation) are secondary outcomes. Innovative translational techniques will be used to provide mechanistic insight, including serum incubation in endothelial cell culture, metabolomics analysis, endothelial cell collections, and assessment of renal blood flow by magnetic resonance imaging. Changes and cerebrovascular and cognitive function will be assessed as part of a sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older; women must be post-menopausal
* Chronic kidney disease stage 3 or 4 (estimated glomerular filtration rate with the 4 CKD-EPI 2021 race-free equation: 20-59 mL/min/1.73m^2; stable renal function in the past 3 months)
* History of inadequately controlled hypertension (systolic blood pressure 120-159 mmHg on two separate days) and on a stable antihypertensive regimen for the past 6 weeks
* Weight stable in the prior 3 months (<2 kg weight change) and willing to remain weight stable throughout the study. Participants using glucagon-like peptide-1 receptor agonists or planning to start them during the study are excluded unless they have achieved weight stability for at least 3 months prior to enrollment.
* Ability to provide informed consent

Exclusion Criteria:

* Patients with advanced chronic kidney disease requiring chronic dialysis
* Significant pulmonary disorders including: chronic obstructive pulmonary disease, interstitial lung disease, cystic fibrosis, or uncontrolled asthma
* History of spontaneous pneumothorax, collapsed lung due to traumatic injury that has not fully healed, burst eardrum that has not fully healed, or other conditions of the eardrum
* Significant co-morbid conditions with a life expectancy of < 1 year
* History of severe congestive heart failure (i.e., ejection fraction <35%)
* History of hospitalization within the last month
* Albuminuria (albumin to creatinine ratio > 2200 mg/g
* Current smoker
* Immunosuppressant agents taken in the past 12 months. Steroids used for the treatment of gout are acceptable; however, patients should not be using steroids within 2 weeks (or 14 days) prior to the vascular testing (rationale: may confound vascular testing)
* Known malignancy
* Inability to cooperate with or clinical contraindication for magnetic resonance imaging including: severe claustrophobia, implants, devices, or non-removable body piercings (these individuals can participate in the study but are excluded from the MRI procedure)
* Illicit drug use or alcohol dependence/abuse, which in the opinion of the investigators, would prohibit compliance with the study intervention

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Casual Systolic Blood Pressure | Baseline, 3 months
  Casual (resting) measures of systolic blood pressure (mmHg) will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure, using an automated oscillometric sphygmomanometer.

SECONDARY OUTCOMES:
Change in 24-Hour Ambulatory Systolic Blood Pressure | Baseline, 3 months
  Brachial artery systolic blood pressure (mmHg) will be measured automatically every 20 minutes for a 24-hour period by an ambulatory blood pressure monitor and will be averaged over the entire 24-hour period.
Change in Brachial Artery Flow-Mediated Dilation | Baseline, 3 months
  Flow-mediated dilation of the brachial artery will be performed using ultrasonography and analyzed with a commercially available software package as percent change in diameter from baseline following reactive hyperemia.

OTHER OUTCOMES:
Change in Ex Vivo Nitric Oxide Production | Baseline, 3 months
  Human umbilical vein and/or cerebral endothelial cells will be incubated with basal media supplemented with 10% human serum collected from participants and stained with the fluorescent probe DAF-FM diacetate to detect nitric oxide production production in response to acetylcholine.
Change in Ex Vivo HUVEC eNOS Activation | Baseline, 3 months
  Human umbilical vein and/or endothelial cells will be treated with 10% human serum and protein expression of cell lysates will be determined by capillary electrophoresis immunoassay.
Change in Ex Vivo Reactive Oxygen Species Production | Baseline, 3 months
  Human umbilical vein endothelial cells will be incubated with basal media supplemented with 10% human serum collected from participants and stained with the fluorescent probe CellROX Deep Red to detect reactive oxygen species production.
Change in Endothelial Cell Protein Expression of MnSOD | Baseline, 3 months
  In a sub-group of participants, endothelial will be obtained from peripheral veins via endovascular biopsy, recovered by centrifugation, fixed, and analyzed for protein expression of MnSOD in collected endothelial cells relative to human umbilical vein endothelial cells using immunofluorescence.
Change in Endothelial Cell Protein Expression of NADPH oxidase | Baseline, 3 months
  In a sub-group of participants, endothelial will be obtained from peripheral veins via endovascular biopsy, recovered by centrifugation, fixed, and analyzed for protein expression of NADPH oxidase in collected endothelial cells relative to human umbilical vein endothelial cells using immunofluorescence.
Change in Endothelial Cell Abundance of Nitrotyrosine | Baseline, 3 months
  In a sub-group of participants, endothelial will be obtained from peripheral veins via endovascular biopsy, recovered by centrifugation, fixed, and analyzed for abundance of nitrotyrosine in collected endothelial cells relative to human umbilical vein endothelial cells using immunofluorescence.
Change in Renal Blood Flow | Baseline, 3 months
  Magnetic resonance imaging will be used to determine flow of the renal arteries.
Adherence | 3 months
  Adherence will be evaluated as percent of completed training sessions at the required workload using data stored on the training device.
Safety (adverse events) | 3 months
  Safety will be evaluated as the number of participants with treatment-related adverse events in each group.
Tolerability (drop-out due to adverse events) | 3 months
  Tolerability will assessed as the rate at which enrolled subjects drop out due to adverse events.
Change in Casual Diastolic Blood Pressure | Baseline, 3 months
  Casual (resting) measures of diastolic blood pressure (mmHg) will be measured in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between each measure, using an automated oscillometric sphygmomanometer.
Change in 24-Hour Ambulatory Diastolic Blood Pressure | Baseline, 3 months
  Brachial artery diastolic blood pressure (mmHg) will be measured automatically every 20 minutes for a 24-hour period by an ambulatory blood pressure monitor and will be averaged over the entire 24-hour period.
Change in Endothelium-Independent Dilation | Baseline, 3 months
  Endothelium-independent dilation will be determined using ultrasonography and analyzed with a commercially available software package as percent chance in brachial artery diameter following 0.4 mg of sublingual nitroglycerin.
Change in middle cerebral artery cerebrovascular reactivity | Baseline, 3 months
  Change in middle cerebral artery velocity in response to hypercapnia
Change in internal carotid artery cerebrovascular reactivity | Baseline, 3 months
  Internal carotid artery diameter in response to hypercapnia
Change in middle cerebral artery pulsatility index | Baseline, 3 months
  Pulsatility index of the middle cerbral artery via transcranial doppler
Change in brain blood flow | Baseline, 3 months
  Total brain blood flow measured via ultrasonography of the internal carotid and vertebral arteries
Change in NIH toolbox cognitive function | Baseline, 3 months
  Total composite score using the NIH toolbox exam
Change in executive function | Baseline, 3 months
  Time to complete the trailmaking test part B

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Nowak, PhD, MPH, Principal Investigator — University of Colorado, Denver; Michel Chonchol, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in CKD. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Oh ES, Opoku G, Darvish S, Craighead DH, Ostrow A, Rossman MJ, Steele CN, Struemph T, You Z, Seals DR, Chonchol M, Nowak KL. Sex Differences in Dementia and Mild Cognitive Impairment in Nondialysis CKD. Clin J Am Soc Nephrol. 2025 Nov 20. doi: 10.2215/CJN.0000000922. Online ahead of print. No abstract available. PMID 41264372
- [Derived] Kistler BM, Kirkman DL, Kusni D, Martin Alemany G, Ribeiro HS, Tarca B, Thompson S, Viana JL, Wilkinson TJ, Wilund KR. Physical Activity and Exercise for Cardiometabolic Health and Fitness in CKD: An Overview by Exercise Type. Clin J Am Soc Nephrol. 2025 Jun 12. doi: 10.2215/CJN.0000000784. Online ahead of print. PMID 40504623